CLINICAL TRIAL: NCT03339687
Title: Research Group RISKDYNAMICS, Sub-Project 8, Work Package 1, Study 2: Addiction Risk: The Influence of Mindset Induction on the Effect of a Brief Intervention to Reduce Alcohol Use
Brief Title: Addiction Risk: The Influence of Mindset Induction on the Effect of a Brief Intervention to Reduce Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Michael Odenwald, Director Outpatient Clinic for Psychotherapy, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OD 113/2-1(2)
Record Dates: First submitted 2017-05-10; First posted 2017-11-13 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction of Open Mindset (Experimental): Psychological Intervention. Participants are asked to work on a brief paper-and-pencil task that has been shown to induce a Deliberative Mindset according to the Mindset theory of action phases (Gollwitzer & Keller (2016). Mindset Theory. In: V. Zeigler-Hill, T.K. Shackelford (eds.), Encyclopedia of Personality and Individual Differences. New York: Springer).
  Interventions: Behavioral: Experimental Mindset Induction
- Induction of a Closed Mindset (Experimental): Psychological Intervention. Participants are asked to work on a brief paper-and-pencil task that has been shown to induce an Implemental Mindset according to the Mindset theory of action phases (Gollwitzer & Keller (2016). Mindset Theory. In: V. Zeigler-Hill, T.K. Shackelford (eds.), Encyclopedia of Personality and Individual Differences. New York: Springer).
  Interventions: Behavioral: Experimental Mindset Induction

INTERVENTIONS:
Behavioral: Experimental Mindset Induction — This induction of a psychological state was extensively studied in cognitive science. Gollwitzer & Keller (2016, p.3): "The deliberative mindset is evoked by asking participants to (a) name an unresolved, important personal problem that is causing rumination but for which they have not made a decision yet and (b) reflect on whether to take action or not. Further, to enhance the depth of reflection, participants are requested to list positive and negative, short- and long-term consequences of both deciding to act and not to act; indicating the probability of the occurrence of each of these consequences is required.
  The implemental mindset is evoked by asking participants to think of a personal project for which they have already made the decision to act but did not initiate any action yet. Subsequently, participants are asked to list the steps necessary for successful goal attainment and to plan out in detail when, where, and how they intend to act on each of these steps."

SUMMARY:
Brief Interventions (BI) based on Motivational Interviewing are effective to reduce alcohol use. In this study the investigators test the hypothesis that that an open Mindset increases the positive effects of BI.

Patients who are newly admitted to the psychotherapy outpatient clinic are routinely screened for risky alcohol use. All patients with risky alcohol use are eligible to the study and all receive the WHO's ASSIST-linked BI.

Participants receive a brief Mindset induction prior to receiving BI. They are are randomly assigned to either the induction of an open or a closed Mindset according to Gollwitzer.

The investigators measure the change in alcohol-related risk perception, treatment motivation and real alcohol drinking.

ELIGIBILITY:
Inclusion Criteria:

* admitted to treatment at psychotherapy outpatient clinic

Exclusion Criteria:

* alcohol use disorder
* substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Individual Risk Perception | The questionnaire assesses the variable related to the week before, i.e. time frame 1 week.
  The participant's self-reported risk of experiencing alcohol-related problems is measured with the self-report measure "Questionnaire for Alcohol-related Risk Perception" (German "Fragebogen zur Alkoholbezogenen Risikowahrnehmung", FAR; Klepper, Odenwald & Rockstroh (2016). Risikowahrnehmung und Alkoholabhängigkeit. SUCHT, 62 (6), 374-382; DOI 10.1024/0939-5911/a000457).

SECONDARY OUTCOMES:
Amount of alcohol drinking | The interviewers assess the number of standard units of alcohol consumed during month before assessment, i.e. time-frame 1 month
  Self-reported amount of standard units of alcohol consumed by the individual

CONTACTS AND LOCATIONS:
Overall Officials: Michael Odenwald, PhD, Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Psychotherapy Outpatient Clinic, Konstanz, Germany

IPD SHARING:
Plan to Share IPD: No